CLINICAL TRIAL: NCT01825031
Title: Reduction of Early mortALITY in HIV-infected African Adults and Children Starting Antiretroviral Therapy: a Randomised Controlled Trial
Brief Title: Reduction of EArly mortaLITY in HIV-infected Adults and Children Starting Antiretroviral Therapy
Acronym: REALITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anna Griffiths, MRC (Other Government)
Collaborators: Department for International Development, United Kingdom (Other Government); Wellcome Trust (Other); Medical Research Council (Other Government); PENTA Foundation (Network)
Responsible Party: Sponsor-Investigator, Anna Griffiths, MRC, Trial Manager, Medical Research Council
Organization: Medical Research Council (Other Government)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ISRCTN43622374
Record Dates: First submitted 2013-01-07; First posted 2013-04-05 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium; Fluconazole; Azithromycin; Albendazole; Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Antiretroviral Therapy (Experimental): Raltegravir twice daily for 12 weeks from antiretroviral therapy (ART) initiation in addition to 3 standard ARVs (2NRTIs/1NNRTI) compared with 3 standard ARVs
  Interventions: Drug: Raltegravir
- Opportunistic Infection (OI) Prophylaxis (Experimental): Immediate isoniazid/pyridoxine and cotrimoxazole, plus 12 weeks fluconazole, 5 days azithromycin and a single dose of albendazole compared with immediate cotrimoxazole (if not already taking this) in all patients plus (not malawi)isoniazid/pyridoxine after 12 weeks.
  Interventions: Drug: Fluconazole; Drug: Azithromycin; Drug: Albendazole; Drug: Isoniazid
- Nutritional Support (Experimental): Supplementation with Ready to Use Supplementary Food (RUSF) for 12 weeks compared with supplementation for those with severe malnutrition as local practice.
  Interventions: Dietary Supplement: Ready to Use Supplementary Food

INTERVENTIONS:
Drug: Raltegravir — 400mg twice daily for the first 12 weeks only in addition to 3 standard ARVs
  Arms: Antiretroviral Therapy
Drug: Fluconazole — 100mg once daily for 12 weeks
  Arms: Opportunistic Infection (OI) Prophylaxis
Drug: Azithromycin — 500mg once daily for 5 days
  Arms: Opportunistic Infection (OI) Prophylaxis
Drug: Albendazole — a single dose 400mg
  Arms: Opportunistic Infection (OI) Prophylaxis
Drug: Isoniazid — 300mg taken immediately in combination with cotrimoxazole
  Arms: Opportunistic Infection (OI) Prophylaxis
Dietary Supplement: Ready to Use Supplementary Food — 2x92g packets daily of high energy, low protein lipid-based paste for 12 weeks
  Other Names: RUSF
  Arms: Nutritional Support

SUMMARY:
A randomised controlled trial to investigate three methods to reduce early mortality in adults, adolescents and children aged 5 years or older starting antiretroviral therapy (ART) with severe immuno-deficiency. The three methods are:

(i) increasing the potency of ART with a 12 week induction period using 4 antiretroviral drugs from 3 classes

(ii) augmented prophylaxis against opportunistic/bacterial infections and helminths for 12 weeks

(iii) macronutrient intervention using ready-to-use supplementary food for 12 weeks.

DETAILED DESCRIPTION:
REALITY is a open-label randomised trial of 1800 adults, adolescents and children aged 5 years or more with low CD4 counts about to initiate ART.

The trial will have a factorial design with 3 randomisations, each to address one of the potential approaches to reduce early mortality in adults and children initiating ART with low CD4, namely:

1. Raltegravir for 12 weeks from ART initiation in addition to 3 standard ART (3-drug 2-class) versus standard of care first-line 3-drug 2-class ART (choice according to national guidelines for ART initiation);
2. Immediate enhanced opportunistic infections (OI) prophylaxis with isoniazid/pyridoxine and cotrimoxazole, plus 12 weeks fluconazole, 5 days azithromycin and a single dose of albendazole versus cotrimoxazole prophylaxis alone for the first 12 weeks followed by isoniazid and any prophylaxis and/or treatment prescribed at screening
3. supplementation with Ready to Use Supplementary Food (RUSF) for 12 weeks versus standard of care nutritional support to those with poor nutritional status according to local guidelines.

All participants will receive cotrimoxazole throughout the trial.

The primary objective of the trial is to identify effective, safe and acceptable interventions to reduce early mortality (all-cause) in HIV-infected adults, adolescents, and older children (5 years or more) initiating ART.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5 years or older
* Documented HIV infection by HIV ELISA or HIV rapid test
* Naive to ART
* CD4 T-cell count <100 cells/mm3 on blood test taken at screening for REALITY
* Results of screening haematology and biochemistry tests available and no contraindications to planned ART according to national guidelines
* Patient/carer provide informed consent (and children <18 years assent, as appropriate according to their age and knowledge of HIV status)

The lower age limit is because CD4 counts are less reliable predictors of immunodeficiency under 5 years: CD4 counts are recommended by guidelines in older children.

No patient with a CD4 count above 100 cells/mm3 should have ART delayed in order to subsequently meet eligibility criteria. Rather, patients eligible for REALITY will be those testing HIV positive for the first time with a low CD4 count (i.e. those delaying presentation to care), or those who have defaulted before initiating ART and only return to care at an advanced stage of immuno-deficiency.

Exclusion Criteria:

* Contraindications to any proposed antiretroviral drugs (including integrase inhibitors), isoniazid, fluconazole, albendazole or azithromycin
* Pregnant or breastfeeding or intending to become pregnant during the first 12 weeks of the study
* Ever known to have previously received single-dose nevirapine for prevention of mother-to-child transmission (mother or child).

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1805 (Actual)
Dates: Start 2013-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
All-cause mortality over the first 24 weeks after starting ART | Week 24

SECONDARY OUTCOMES:
48 week mortality (all-cause) | Week 48
Safety | Week 0-48
  * serious adverse events
  * grade 4 adverse events
  * adverse events leading to modification of ART or other study drugs
Hospital inpatient episodes and total days admitted | Week 0-48
Adherence to ART and acceptability of each strategy | Week 0-48
  Adherence to ART, OI drugs and RUSF will be assessed in all participants at each visit by pill counts and short nurse-administered questions. Every 12 weeks, a more detailed adherence questionnaire will be adminstered.
Endpoint relating to anti-infection intervention | 0-48 weeks
  Incidence of tuberculosis (TB), cryptococcal and candida disease, severe bacterial infections
Endpoint relating to anti-malnutrition intervention | 0-48 weeks
  BMI, weight and body fat assessed by bioimpedance analysis (BIA), height (in children) and grip strength
Endpoint relating to anti-HIV intervention | 0-48 weeks
  Changes in CD4 cell count

CONTACTS AND LOCATIONS:
Overall Officials: Diana M Gibb, Study Director — Medical Research Council
Locations (8):
- Kenya (2):
  - Moi University Clinical Research Centre, Eldoret
  - KEMRI Wellcome Trust Research Programme, Kilifi
- University of Malawi, Blantyre, Malawi
- Uganda (4):
  - Joint Clinical Research Centre, Fort Portal, Fort Portal
  - Joint Clinical Research Centre, Gulu, Gulu
  - Joint Clinical Research Centre, Mbale, Mbale
  - Joint Clinical Research Centre, Mbarara, Mbarara
- University of Zimbabwe Clinical Research Centre, Harare, Zimbabwe

REFERENCES:
- [Derived] Kelly C, Tinago W, Alber D, Hunter P, Luckhurst N, Connolly J, Arrigoni F, Garcia Abner A, Kamn'gona R, Sheha I, Chammudzi M, Jambo K, Mallewa J, Rapala A, Mallon PWG, Mwandumba H, Klein N, Khoo S. Inflammatory pathways amongst people living with HIV in Malawi differ according to socioeconomic status. PLoS One. 2021 Aug 25;16(8):e0256576. doi: 10.1371/journal.pone.0256576. eCollection 2021. PMID 34432828
- [Derived] Kelly C, Tinago W, Alber D, Hunter P, Luckhurst N, Connolly J, Arrigoni F, Abner AG, Kamngona R, Sheha I, Chammudzi M, Jambo K, Mallewa J, Rapala A, Heyderman RS, Mallon PWG, Mwandumba H, Walker AS, Klein N, Khoo S. Inflammatory Phenotypes Predict Changes in Arterial Stiffness Following Antiretroviral Therapy Initiation. Clin Infect Dis. 2020 Dec 3;71(9):2389-2397. doi: 10.1093/cid/ciaa186. PMID 32103268
- [Derived] Kityo C, Szubert AJ, Siika A, Heyderman R, Bwakura-Dangarembizi M, Lugemwa A, Mwaringa S, Griffiths A, Nkanya I, Kabahenda S, Wachira S, Musoro G, Rajapakse C, Etyang T, Abach J, Spyer MJ, Wavamunno P, Nyondo-Mipando L, Chidziva E, Nathoo K, Klein N, Hakim J, Gibb DM, Walker AS, Pett SL; REALITY trial team. Raltegravir-intensified initial antiretroviral therapy in advanced HIV disease in Africa: A randomised controlled trial. PLoS Med. 2018 Dec 4;15(12):e1002706. doi: 10.1371/journal.pmed.1002706. eCollection 2018 Dec. PMID 30513108
- [Derived] Mallewa J, Szubert AJ, Mugyenyi P, Chidziva E, Thomason MJ, Chepkorir P, Abongomera G, Baleeta K, Etyang A, Warambwa C, Melly B, Mudzingwa S, Kelly C, Agutu C, Wilkes H, Nkomani S, Musiime V, Lugemwa A, Pett SL, Bwakura-Dangarembizi M, Prendergast AJ, Gibb DM, Walker AS, Berkley JA; REALITY trial team. Effect of ready-to-use supplementary food on mortality in severely immunocompromised HIV-infected individuals in Africa initiating antiretroviral therapy (REALITY): an open-label, parallel-group, randomised controlled trial. Lancet HIV. 2018 May;5(5):e231-e240. doi: 10.1016/S2352-3018(18)30038-9. Epub 2018 Apr 10. PMID 29653915